CLINICAL TRIAL: NCT04215120
Title: A Phase 3, Multicenter, Open-label, Randomized, Active-controlled Study to Evaluate the Efficacy and Safety of Desidustat Tablet Versus Epoetin Alfa Injection for the Treatment of Anemia in Patients With Chronic Kidney Disease (CKD) on Dialysis (DREAM-D)
Brief Title: Desidustat in the Treatment of Anemia in CKD on Dialysis Patients
Acronym: DREAM-D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DESI.19.001.01
Record Dates: First submitted 2019-12-22; First posted 2020-01-02 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-01

CONDITIONS: Chronic Kidney Disease Stage 5 on Dialysis
MeSH Terms: interventions — desidustat; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desidustat oral tablet (Active Comparator): Randomly assigned to receive Desidustat 100 mg in a 1:1 ratio for 24 weeks.
  Interventions: Drug: Desidustat Oral Tablet
- Epoetin Injection (Experimental): Randomly assigned to receive Epoetin in a 1:1 ratio for 24 weeks.
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: Desidustat Oral Tablet — Desidustat tablet
  Arms: Desidustat oral tablet
Drug: Epoetin Alfa — Epoetin Injection
  Arms: Epoetin Injection

SUMMARY:
A phase 3, multicenter, open-label, randomized, active-controlled study to evaluate the efficacy and safety of Desidustat Tablet versus Epoetin alfa Injection for the treatment of anemia in patients with CKD on dialysis. (DREAM-D)

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and give informed consent for participation. 2. Hemoglobin values during the screening period must be 8-11 g/dL (both inclusive).

3.

1. Patients will be considered not treated with erythropoietin analogue (Epoetin and Darbepoeitin) if they have not received erythropoietin analogue for at least 4 weeks and Mircera® for at least 8 weeks prior to screening visit. OR
2. Patients who are on ESA therapy must be on stable dose for 4 weeks prior to enrollment (≤30% of dose change).

   4. Patients on hemodialysis (≥2 times in a week) for at least 12 weeks prior to screening visit and have access consisting of an arteriovenous fistula, AV graft, or catheter (permanent/temporary).

   5. Patients with no planned change in dialysis modality and with no planned renal transplant during study period.

   6. Left ventricular ejection fraction ≥40% by echocardiogram prior to randomization.

   7. No iron, folate or Vitamin B12 deficiency.

   8. Females of childbearing potential, must agree to use one of the approved contraception methods, from screening until completion of the follow-up visit.

   Exclusion Criteria:
   1. Red blood cell transfusion within 8 weeks prior to participating in the study.
   2. History of previous or concurrent cancer.
   3. Serologic status reflecting active hepatitis B or C infection or Human immunodeficiency virus (HIV) infection.
   4. Active infection at initiation of study.
   5. History of renal transplant.
   6. Uncontrolled hypertension (defined as SBP >180 mmHg or DBP >100 mmHg) at screening visit (before dialysis).
   7. Patient on high rhEPO dose at screening visit. [High dose defined as an epoetin dose of ≥450 IU/kg/week intravenous or ≥ 300 IU/kg/week subcutaneous or darbepoetin dose of ≥1.5 µg/kg/week subcutaneous].
   8. Major surgery within 90 days of the first day of study drug dosing, and minor surgery within 30 days of the first day of study drug dosing.
   9. Unable to swallow tablets or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption such as; malabsorption syndrome, resection of the small bowel or poorly controlled inflammatory bowel disease affecting the small intestine.
   10. History of uncontrolled autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura (ITP) or thalassemia.
   11. Presence or a history of bleeding disorders or clinical conditions (e.g. gastrointestinal [GI] bleeding or constitutional disorders) that may increase risk of life-threatening bleeding.
   12. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
   13. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Desidustat or Epoetin alfa or to any erythropoieisis-stimulating agent.
   14. Pregnant and breastfeeding women.
   15. Current life-threatening illness, medical condition or organ system dysfunction which, in the Investigator's opinion, could compromise the patient's safety.
   16. Other laboratory abnormalities that, in the opinion of the investigator, would compromise the patient's safety or interfere with data interpretation.
   17. Presence of other clinically significant systemic disorders or diseases (e.g., respiratory, gastrointestinal, endocrine, immunological, dermatological, neurological, psychiatric disease or any other body system involvement) which, in the Investigator's opinion, could compromise the patient's safety.
   18. History of significant alcoholism or drug abuse within the past 1 year. History or presence of significant smoking (more than 10 cigarettes per day) or consumption of tobacco/nicotine products (more than 10 times per day).
   19. History of difficulty with donating blood.
   20. History or presence of any clinically significant electrocardiogram (ECG) abnormalities during screening.
   21. Participants who have participated in any drug research study other than the present trial within past 3 months.
   22. Participants who have donated one unit (350 ml) of blood in the past 3 months or history of whole blood transfusion in last 120 days prior to entry in the study.
   23. Existing clinically active chronic inflammatory disease (RA, Celiac disease, UC, Crohns disease)
   24. In case of DM patients, HbA1c >9%.
   25. Female volunteers with following criteria will not be recruited:

       * History of pregnancy or lactation in the past 3 months
       * Fertile female volunteers not protected against pregnancy by adequate long- term anti-fertility measures
       * History of less than 1 year of menopause and not using adequate long-term anti-fertility measures
       * Positive urine pregnancy test at Visit 2
       * Positive serum β-hCG level at the screening visit
   26. Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification or history of myocardial infarction prior to first dose with study drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | 24 weeks
  Change in Hb levels from baseline

SECONDARY OUTCOMES:
Hemoglobin Response | 24 weeks
  No. of subjects with Hb response
Hemoglobin target range | 24 weeks
  Time to achieve target range Hb level

CONTACTS AND LOCATIONS:
Overall Officials: Dr Deven Parmar, MD, Study Director — Zydus Lifesciences Limited
Locations (7):
- India (7):
  - Karnavati Hospital Pvt.Ltd, Ahmedabad, Gujarat
  - Shalby Hospital,, Ahmedabad, Gujarat
  - DHS Multispecialty Hospital, Ahmedabad, Gujarat
  - Chopda Medicare & Research Centre Pvt. Ltd, Nashik, Maharashtra
  - Aditya Birla Memorial Hospital, Pune, Maharashtra
  - Eternal Hospital, Jaipur, Rajasthan
  - Star Hospital, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278